CLINICAL TRIAL: NCT00786019
Title: Influence Of Endothelial Function On Central and Peripheral Causes Of Exercise Impairment In Type 2 Diabetes
Acronym: InsITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Diabetes Association (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 07-1152; UL1TR000154 (NIH)
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Results first posted 2018-09-11 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Type 2 Diabetes
Keywords: Type; 2; Diabetes; Blood; Vessel; Function; Exercise; Program; Intervention; Vitamin; C; Men; Women; Blood vessel function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Limb-girdle muscular dystrophy, type 2C; Diabetes Mellitus; Motor Activity; Multiple Endocrine Neoplasia Type 1 | interventions — Resistance Training; Exercise; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ascorbic acid (Experimental): All study subjects have ascorbic acid infusion during one exercise visit as well as a three month exercise training intervention.
  Interventions: Behavioral: Exercise program; Drug: Ascorbic Acid (Vitamin C)

INTERVENTIONS:
Behavioral: Exercise program — Three month exercise program located at the Anschutz Medical Campus at I-225 and Colfax. The program runs three times per week for about an hour each session. Gym is open Monday - Saturday during specific hours (morning, noon, evening).
  Other Names: Exercise Training
Drug: Ascorbic Acid (Vitamin C) — During one exercise study visit, 0.06 grams of Vitamin C per kilogram fat-free mass per 100 milliliters (mL) of normal saline administered; Subjects will receive a bolus of 100mL Vitamin C solution given at 5ml/minute over 20 minutes followed by a "drip-infusion" given at 1.7ml/minute.
  Other Names: Ascorbic Acid; Vitamin C

SUMMARY:
This study will evaluate the effects of impaired blood flow regulation on exercise. It will also determine whether the effects are more important in the heart or in the skeletal muscle tissue during exercise. In addition, this study will decide whether temporarily reversing these problems will improve blood flow control, improve heart and muscle tissue function and help improve exercise capacity in person with type 2 diabetes. This study will do so using two methods: (1) by giving vitamin C intravenously (IV) and (2) a three month exercise training program. Up to 100 subjects will be enrolled in this study.

DETAILED DESCRIPTION:
The investigators have found that persons with type 2 diabetes have an impaired ability to perform exercise even without clinically apparent complications. The reasons for this marked abnormality are unknown but are important as the decreased ability to exercise could contribute to the decreased expenditure of physical activity frequently observed in this population and may potentially constitute an early marker of cardiovascular disease.

The investigators wish to evaluate the effects of impaired blood flow regulation on exercise capacity and whether the effects are more important in the heart or in the skeletal muscle tissue during exercise. In addition, the investigators are determining whether correcting these abnormalities by two methods of improving blood flow regulation (acutely infusing Vitamin C or three months of chronic exercise training) leads to improved blood flow regulation, improved heart and skeletal muscle tissue function and hence to better exercise capacity in person with type 2 diabetes. This information will provide a more mechanistic understanding of causes of abnormal exercise responses observed in person with type 2 diabetes as well as whether and to what degree responses are modifiable. Interventions that reverse the exercise defect may facilitate patient adherence to prescribed physical activity programs and potentially decrease cardiovascular mortality in this large segment of the population.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with uncomplicated Type 2 Diabetes
* Healthy men and women without Type 2 Diabetes
* Patients with Type 2 Diabetes may be taking metformin or sulfonylurea drugs to treat diabetes
* Persons with history of hypercholesteremia if controlled with statins and/or diet
* Patients who are moderately overweight (BMI 25-37.5)
* Must be sedentary (defined as regular exercise < 2 times a week at a low to moderate level).
* Patients with Hemoglobin A1c (HBA1C) <8%
* Patients between the ages of 30 to 55 years
* Premenopausal women.
* Former smokers who have quit smoking for at least one year
* Absence of comorbid conditions
* Mild neuropathy is O.K. as long as it will not hamper exercise performance.
* Resting systolic blood pressure (SBP) < 140, Resting diastolic blood pressure (DBP) < 90
* Total Cholesterol < 205 Triglycerides < 250 low density lipoprotein (LDL) < 130
* Control subjects with a normal A1C and fasting glucose

Exclusion Criteria:

* People with T2DM taking oral medications, other than metformin or sulfonylurea drugs to control their diabetes.
* Persons treated with insulin will be excluded
* People who are currently smoking or have not quit for at least one year
* Controls who have immediate family history of T2DM
* Peri-menopausal or post-menopausal women.
* Peripheral neuropathy
* Total cholesterol > 205
* Regional wall motion abnormalities
* LV wall thickness ≥1.1 cm
* Decreased contractility (fractional shortening <30%)
* Ischemic heart disease (abnormal resting or exercise ECG)
* Presence of angina that would limit exercise performance
* Pulmonary problems that would limit exercise performance
* Systolic blood pressure >140 mmHg at rest or >250 mmHg with exercise or diastolic pressure >90 mmHg at rest or >105 mmHg with exercise
* Persons with autonomic insufficiency, assessed by measuring variation in RR intervals with cycled breathing and by presence of a >20 mm fall in upright blood pressure without a change in heart rate
* Proteinuria (urine protein >200 mg/dl) or a creatinine > 2 mg/dl
* Renal disease

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2008-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith G Regensteiner, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Scalzo RL, Bauer TA, Harrall K, Moreau K, Ozemek C, Herlache L, McMillin S, Huebschmann AG, Dorosz J, Reusch JEB, Regensteiner JG. Acute vitamin C improves cardiac function, not exercise capacity, in adults with type 2 diabetes. Diabetol Metab Syndr. 2018 Feb 14;10:7. doi: 10.1186/s13098-018-0306-9. eCollection 2018. PMID 29456629

RESULTS

PARTICIPANT FLOW:
Groups:
- Ascorbic Acid - Control: All study subjects have ascorbic acid infusion during one exercise visit as well as a three month exercise training intervention.
  Exercise program: Three month exercise program located at the Anschutz Medical Campus. The program runs three times per week for about an hour each session.
  Ascorbic Acid (Vitamin C): During one exercise study visit, 0.06 grams of Vitamin C per kilogram (kg) fat-free mass per 100 milliliters (mL) of normal saline administered; Subjects will receive a bolus of 100mL Vitamin C solution given at 5ml/minute over 20 minutes followed by a "drip-infusion" given at 1.7ml/minute.
- Ascorbic Acid - Type 2 Diabetes: All study subjects have ascorbic acid infusion during one exercise visit as well as a three month exercise training intervention.
  Exercise program: Three month exercise program located at the Anschutz Medical Campus. The program runs three times per week for about an hour each session.
  Ascorbic Acid (Vitamin C): During one exercise study visit, 0.06 grams Vitamin C per kilogram fat-free mass per 100 milliliters (mL) of normal saline administered; Subjects will receive a bolus of 100mL Vitamin C solution given at 5ml/minute over 20 minutes followed by a "drip-infusion" given at 1.7ml/minute.
Period: Overall Study
Arm/Group | Ascorbic Acid - Control | Ascorbic Acid - Type 2 Diabetes
Started | 20 | 27
Completed | 15 | 17
Not Completed | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Ascorbic Acid - Type 2 Diabetes: All study subjects have ascorbic acid infusion during one exercise visit as well as a three month exercise training intervention.
  Exercise program: Three month exercise program located at the Anschutz Medical Campus. The program runs three times per week for about an hour each session.
  Ascorbic Acid (Vitamin C): During one exercise study visit, 0.06 grams of Vitamin C per kilogram (kg) fat-free mass per 100 milliliters (mL) of normal saline administered; Subjects will receive a bolus of 100mL Vitamin C solution given at 5ml/minute over 20 minutes followed by a "drip-infusion" given at 1.7ml/minute.
- Total: Total of all reporting groups
Arm/Group | Ascorbic Acid - Control | Ascorbic Acid - Type 2 Diabetes | Total
Number analyzed (Participants) | 20 | 27 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (6.0) | 46.5 (5.7) | 46.0 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 9 | 21 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 2 | 2
  Black/African American | 6 | 7 | 13
  Hispanic | 4 | 5 | 9
  White | 10 | 11 | 21
  American Indian | 0 | 1 | 1
  Other | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 27 | 47
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 171.30 (10.8) | 175.17 (8.7) | 173.52 (9.7)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 89.67 (10.8) | 97.89 (18.0) | 94.39 (15.8)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.60 (3.0) | 31.75 (4.7) | 31.26 (4.0)
Body Fat Percentage (%) [Mean (Standard Deviation); unit: percentage] | 35.00 (7.0) | 32.61 (6.1) | 33.63 (6.5)
Glucose (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 87.15 (5.7) | 118.33 (22.2) | 105.06 (23.1)
Insulin (uIU/mL) [Mean (Standard Deviation); unit: uIU/mL] | 15.45 (7.7) | 29.93 (19.6) | 23.77 (17.1)
Total Cholesterol (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 173.45 (28.8) | 147.30 (20.6) | 158.43 (27.5)
Triglycerides (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 108.55 (37.1) | 151.52 (65.5) | 133.23 (58.8)
LDL Cholesterol (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 105.00 (22.4) | 87.33 (19.2) | 94.85 (22.2)
HDL Cholesterol (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 52.2 (13.0) | 38.26 (8.1) | 44.19 (12.5)
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage] | 5.37 (0.4) | 6.85 (0.7) | 6.22 (1.0)
Peak VO2 (relative) [Mean (Standard Deviation); unit: mL/kg/min] | 22.32 (4.9) | 20.93 (3.8) | 21.52 (4.3)
Peak VO2 (absolute) [Mean (Standard Deviation); unit: mL/min] | 2027.65 (529.2) | 2076.67 (531.6) | 2055.81 (525.3)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Circumferential Strain Before and After Exercise at Baseline, After Vitamin C Infusion, and After Exercise Training
Description: Characterize the purported cardiac dysfunction during exercise in people with type 2 diabetes (T2D). In a normal patient when measuring circumferential strain, results are negative with downward tracing (as strain is a relative change in length). Circumferential strain is a measurement of ventricular circumference within the heart vessels, measured via echocardiography.
Time Frame: 7 months; Measures are made at rest and after exercise for baseline, at rest and after infusion for Vitamin C administration, and at rest and after exercise following the exercise training
Measure: Mean (Standard Deviation); unit: percentage of change in length
Groups:
- Circumferential Strain - Control; Circumferential Strain - Type 2 Diabetes: All study subjects have ascorbic acid infusion during one exercise visit as well as a three month exercise training intervention.
  Exercise program: Three month exercise program located at the Anschutz Medical Campus. The program runs three times per week for about an hour each session.
  Ascorbic Acid (Vitamin C): During one exercise study visit, 0.06 grams of Vitamin C per kilogram (kg) fat-free mass per 100 milliliters (mL) of normal saline administered; Subjects will receive a bolus of 100mL Vitamin C solution given at 5ml/minute over 20 minutes followed by a "drip-infusion" given at 1.7ml/minute.
Arm/Group | Circumferential Strain - Control | Circumferential Strain - Type 2 Diabetes
Number analyzed (Participants) | 15 | 17
percentage of change in length
  Baseline | -24 (1) | -20 (1)
  Vitamin C | -23 (1) | -21 (1)
  Post Exercise Training | -22 (1) | -22 (1)

2. Primary Outcome: Ejection Fraction: Percentage of Blood Leaving the Heart Before and After Exercise at Baseline, After a Vitamin C Infusion, and After Exercise Training
Description: Evaluate potential changes in cardiac function by echocardiography following 2 interventions: Three months of exercise training and acute vitamin C administration. Ejection fraction (EF) is a measurement of the percentage of blood leaving your heart each time it contracts, typically measure by echocardiography. Numbers listed are absolute EF values.
Time Frame: 7 months; Measures are made at rest for baseline, at rest for Vitamin C administration, and at rest following the exercise training
Measure: Mean (Standard Deviation); unit: percentage of blood leaving the heart
Groups:
- Ejection Fraction - Control; Ejection Fraction - Type 2 Diabetes: All study subjects have ascorbic acid infusion during one exercise visit as well as a three month exercise training intervention.
  Exercise program: Three month exercise program located at the Anschutz Medical Campus. The program runs three times per week for about an hour each session.
  Ascorbic Acid (Vitamin C): During one exercise study visit, 0.06 grams of Vitamin C per kilogram (kg) fat-free mass per 100 milliliters (mL) of normal saline administered; Subjects will receive a bolus of 100mL Vitamin C solution given at 5ml/minute over 20 minutes followed by a "drip-infusion" given at 1.7ml/minute.
Arm/Group | Ejection Fraction - Control | Ejection Fraction - Type 2 Diabetes
Number analyzed (Participants) | 15 | 17
percentage of blood leaving the heart
  Baseline | 65 (2) | 65 (1)
  Vitamin C | 67 (2) | 63 (1)
  Post Exercise Training | 61 (3) | 65 (3)

ADVERSE EVENTS:
Groups:
- Ascorbic Acid - Control; Ascorbic Acid - T2D: All study subjects have ascorbic acid infusion during one exercise visit as well as a three month exercise training intervention.
  Exercise program: Three month exercise program located at the Anschutz Medical Campus. The program runs three times per week for about an hour each session.
  Ascorbic Acid (Vitamin C): During one exercise study visit, 0.06 g Vit C per kg fat-free mass per 100 ml of normal saline administered; Subjects will receive a bolus of 100mL Vit C solution given at 5ml/min over 20minutes followed by a "drip-infusion" given at 1.7ml/min.
Arm/Group | Ascorbic Acid - Control | Ascorbic Acid - T2D
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/27
Other Adverse Events (participants affected / at risk) | 0/20 | 2/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ascorbic Acid - Control (N=20) | Ascorbic Acid - T2D (N=27)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 — A subject informed study staff that she was pregnant and was immediately withdrawn from the study as per exclusion criteria. A negative pregnancy test was recorded at start of study involvement.
Needle stick (Injury, poisoning and procedural complications) | 0 | 1 — Nursing staff member stuck by participant's used lancet as they were experiencing a feeling of faintness after exercise. Nurse informed HR and visited infectious disease department for testing, all of which was negative.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ascorbic Acid - Control (N=20) | Ascorbic Acid - T2D (N=27)
Vasovagal Episodes (Cardiac disorders) | 0 | 1 — Subject had two vasovagal episodes during initial visits. MD present had no concern; cardiologist found no evidence of ischemia on EKG. Another during intervention, upon which subject was withdrawn from study (pending resolution of health issues).
Minor Exercise Injury (Musculoskeletal and connective tissue disorders) | 0 | 1 — Subject felt pop in L hamstring when on leg curl machine during 7th week of intervention. MD immediately evaluated, advised subject to massage, heat/ice, and take ibuprofen as needed. Next day, no visible swelling, pain substantially reduced.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No